CLINICAL TRIAL: NCT03677076
Title: Clonal Emergence and Regression During Radium-223 Therapy for Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 102691; IIR-US-2017-4183 (Other: Bayer)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary/Correlative: Patients will complete questionnaires and have research blood drawn.
  Interventions: Other: Ancillary/Correlative

INTERVENTIONS:
Other: Ancillary/Correlative — Collection of research blood and urine

SUMMARY:
This study is for patients with metastatic prostate cancer receiving radium-223 as their standard of care therapy. The researchers will collect blood and urine samples from patients before, during and after the radium-223 therapy. The researchers will compare these samples to observe how the treatment has affected different cancer markers.

DETAILED DESCRIPTION:
This study proposes to document the presence of clonal emergence and regression during radium-223 therapy for metastatic prostate cancer by serial ctDNA analysis of tumor-associated mutations, using the clinically-available Guardant 360 platform. These data may provide important mechanistic insights into radium-223 therapy by 1) identifying mutations associated with radium-223 resistance or sensitivity, 2) providing new markers of treatment response in an individual, and 3) revealing antitumor effects from radium-223 that are not easily recognized with standard tumor response metrics. Positive finding based on this clinically-available platform will be readily applied by the oncology treatment community.

ELIGIBILITY:
INCLUSION CRITERIA

1. Prostate adenocarcinoma by history or medical records.
2. Two or more bone metastases as demonstrated by imaging studies (technetium bone scan, fluoride PET scan, FDG PET scan, fluciclovine PET scan, CT scan, or MRI scan) or by biopsy.
3. Patients must be on ADT with a GnRH receptor agonist/antagonist or orchiectomy, with or without an anti-androgen or testosterone synthesis inhibitor. Patients must have a documented castrate level of testosterone (<50ng/dL) and be willing to continue their GnRH agonist/antagonist during the course of radium-223 therapy.
4. Patients may have had localized external beam radiation to as much as 20% of the skeleton
5. Adequate hematopoietic, renal, and hepatic function. These parameters include:

   * Hemoglobin ≥ 10gm/dL
   * WBC ≥ 3.0K/mcL
   * ANC ≥ 1.5K/mcL
   * Platelet count ≥ 100K/mcL
   * Creatinine < 1.5 ng/mL
   * Total bilirubin <1.5 ng/mL.
   * Albumin > 25 g/L
6. Patients should have an elevated, relevant tumor marker such as PSA, CEA, or LDH.
7. Age ≥18 years old
8. Life expectancy of at least 24 weeks
9. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedures. Subjects must be willing and able to comply with the protocol, including follow-up visits and examinations.
10. Men of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent until at least 30 days after the last dose of radium-223 treatment or during the course of radium-223 treatment.
11. Subjects must have had a Guardant 360 ctDNA-based genomic profile performed up to four months prior to the first dose of radium-223, with no new therapy started in the interim. This assay must show at least one single nucleotide variant, either missense or synonymous, or one amplification.
12. Subjects should continue any previously-started bone-hardening agents (zoledronic acid or denosumab) during radium-223 therapy.
13. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v 5.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF).

EXCLUSION CRITERIA

1. Initiation of any additional anti-tumor therapy within 2 months of starting radium-223 treatment
2. Presence of only lytic bone metastases
3. Prior cytotoxic chemotherapy for metastatic PCa
4. Prior systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Radium Ra 223 dichloride) for the treatment of bony metastases
5. Other malignancy requiring systemic therapy within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer)
6. Visceral (i.e. liver, lung, brain, adrenal, brain, but not lymph node) metastases as assessed by chest, abdominal, or pelvic computed tomography, or other imaging modality)
7. Lymphadenopathy exceeding 6 cm in short-axis diameter, or any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis
8. Imminent spinal cord compression based on clinical findings and/or MRI. Treatment should be completed for spinal cord compression.
9. Any infection ≥ Grade 2 per NCI-CTCAE version 5.0
10. Cardiac failure NYHA III or IV
11. Crohn's disease or ulcerative colitis
12. Bone marrow dysplasia, myelodysplasia
13. Fecal incontinence
14. Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
15. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
16. Concurrent use of abiraterone or enzalutamide. A 28-day washout period is required for both agents.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult males with prostate cancer receiving radium223 treatment
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Minor allele frequency (MAF) in ctDNA | 24 months
  The primary objective is to estimate average change in MAF in one or more clonal SNVs, comparing baseline to on-treatment, and baseline to post-treatment samples

SECONDARY OUTCOMES:
Changes in MAF of clonal SNV | 24 months
  • Determine if changes from baseline in MAF of clonal SNVs during therapy and post-treatment differ significantly from 0.
Change in clonal mutation MAF and change in pain | 24 months
  • Evaluate the association between change from baseline in clonal mutation MAF and change in pain (evaluated by VAS pain score and analgesic usage diary), measured both during therapy and post-treatment.
Change in clonal mutation MAF and change in tumor markers | 24 months
  • Evaluate the association between change in clonal mutation MAF and change in tumor markers, including prostate specific antigen (PSA), CEA and LDH, measured by standard biochemical assays both during therapy and post-treatment.
Change in clonal mutation MAF and markers of bone metabolism | 24 months
  • Evaluate the association between change in clonal mutation MAF and markers of bone metabolism including urine N-telopeptide and serum bone-specific alkaline phosphatase, measured by ELISA assays both during therapy and post-treatment.
Change in clonal mutation MAF and presence of the TMPRSS2-ERG fusion gene | 24 months
  • Evaluate the association between change in clonal mutation MAF and presence of the TMPRSS2-ERG fusion gene, measured in plasma/urine by digital PCR Evaluate the association between change in clonal mutation MAF and clinical benefit, (time from the last dose of radium-223 to the initiation of a new systemic therapy, measured at least 60 days after final dose) and change in QOL (measured by FACT-P instrument).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No